CLINICAL TRIAL: NCT06278285
Title: Effect of Agonist GLP1 on Adipose Tissue in Patients Undergoing Bariatric Surgery
Acronym: Maigrir_OT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-AOIP-01
Record Dates: First submitted 2024-02-09; First posted 2024-02-26 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole blood in a GLP1 (Other): Oxytocyne assay in a GLP1 analogue or non-analogue patient population
  Interventions: Other: Blood GLP1
- whole blood in non analague patient population (Other): Oxytocyne assay in a GLP1 analogue or non-analogue patient population
  Interventions: Other: Blood No treated GLP1

INTERVENTIONS:
Other: Blood GLP1 — On the day of surgery, the surgeon will remove visceral adipose tissue (1 cm3) from the operative waste. The adipose tissue is separated into 2 samples, one frozen in nitrogen, the other embedded in formalin. The samples are then sent to the Institut de Biologie de Valrose (iBV) to assess any differences between the two groups of patients (patients treated with anti-GLP-1 analogues
  Arms: whole blood in a GLP1
Other: Blood No treated GLP1 — On the day of surgery, the surgeon will remove visceral adipose tissue (1 cm3) from the operative waste. The adipose tissue is separated into 2 samples, one frozen in nitrogen, the other embedded in formalin. The samples are then sent to the Institut de Biologie de Valrose (iBV) to assess any differences between the two groups of patients (patients treated with patients not treated with anti-GLP-1 analogues) and the presence of fibrosis.
  Arms: whole blood in non analague patient population

SUMMARY:
Normalizing weight gain and preventing the redistribution of body fat is a major health issue, and could help prevent the onset of various symptoms of metabolic syndrome. Above all, it is important to understand the mechanisms by which these different treatments affect adipose tissue. To this end, the investigators will first study the impact of GLP-1 analogues on adipose tissue. The main objective is to show that subjects treated with a GLP-1 agonist have a significant change in their oxytocin levels compared with subjects not treated with a GLP-1 agonist.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age.
* Patient able to read and understand the information/consent leaflet.
* Patient with BMI > 35 with at least one comorbidity. Or BMI > 40
* Indication for digestive surgery validated in a multidisciplinary consultation meeting and prior agreement accepted by the CPAM.
* Membership of a social security scheme
* Patient's signed informed consent
* For subjects in the GLP-1 analogue group: GLP-1 analogue taken for at least 3 months.
* For non-GLP-1 analogue group: never taken GLP-1 analogues.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Vulnerable patients (under guardianship)
* Patients deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-09-06 (Estimated); Study Completion 2027-03-06 (Estimated)

PRIMARY OUTCOMES:
Rate of oxytocin | one time (before surgery)
  show that subjects treated with a GLP-1 agonist have a significant change in oxytocin levels compared with subjects not treated with a GLP-1 agonist.

SECONDARY OUTCOMES:
Fibrosis rate | At surgery
  compare adipose tissue caracteristics between patients treated by analog GLP1 and not treated by analog GLP1

CONTACTS AND LOCATIONS:
Overall Officials: Iannelli Antonio, PhD, Principal Investigator — Clinique Parc Impérial, Service de Chirurgie Digestive
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No